CLINICAL TRIAL: NCT05155046
Title: Phase II Trial of 18F-DCFPyL Imaging as a Method to Assess Treatment Response to Stereotactic Body Radiation Therapy
Brief Title: 18F-DCFPyL Imaging as a Method to Assess Treatment Response to Stereotactic Body Radiation Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000481; 000481-C
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07-16

CONDITIONS: Localized Prostate Cancer
Keywords: Localized Prostate Cancer; Radiotherapy; Prostate Specific Membrane Antigen; Androgen Deprivation Therapy; longitudinal quality of life
MeSH Terms: interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL imaging (Experimental): 18F-DCFPyL imaging with routine imaging (mpMRI)
  Interventions: Drug: 18F-DCFPyL

INTERVENTIONS:
Drug: 18F-DCFPyL — 18F-DCFPyL imaging will be performed at baseline, 8 weeks after ADT initiation, 6 months post SBRT and at recurrence. The target administered activity will be 6.5 mCi with a lower limit of 6 mCi.

SUMMARY:
Background:

Identifying medium- and high-risk prostate cancer early may allow for treatments to work. But identification can be hard. Researchers want to see if a radiotracer used during PET scans can help.

Objective:

To test how an imaging agent called 18F-DCFPyL detects response to standard prostate cancer treatment.

Eligibility:

People ages 18 and older with newly diagnosed prostate cancer who have no evidence of distant metastatic disease and plan to get stereotactic body radiation therapy (SBRT) with or without androgen deprivation therapy (ADT).

Design:

Participants will be screened with:

Medical history

Physical exam

Blood tests

MRI

Participants will have baseline MRI and PET/CT scans. For the MRI, they may get a contrast agent by IV injection. For the PET/CT scan, they will get an IV injection of 18FDCFPyL. About 1 to 2 hours later, they will get the PET/CT scan. During the scans, participants will lie on their back and remain still for 45 minutes to 1 hour. These scans will be repeated at different points during the study.

Participants will get SBRT with or without ADT.

Participants will complete questionnaires about their quality of life.

Participants will be asked about any symptoms they are having. They will also be asked about medications they are using. They may have a physical exam.

Participants will give blood and urine samples. They will give a tumor sample from a biopsy they have had in the past.

After treatment, participants will have follow-up visits. These will occur 1 month after treatment, then every 3 months for a year, and then every 6 months for 1 more year.

DETAILED DESCRIPTION:
Background:

Radiotherapy is a highly effective treatment for localized prostate cancer; however, recurrence is more common in patients with unfavorable intermediate and high-risk prostate cancer, and is usually diagnosed by rising prostate specific antigen (PSA - biochemical failure).

Early identification of disease persistence or recurrence before meeting criteria of biochemical failure may allow effective potentially curative salvage treatment, but identification of local recurrence or persistence at early stages is challenging. CT imaging is relatively insensitive at localizing recurrence, while MRI is more sensitive for local recurrence but is non-specific.

Prostate specific membrane antigen (PSMA) targeted PET imaging was recently FDA approved for imaging men with suspected prostate cancer metastases who are potentially curable by radiation or surgery. PSMA based imaging has been used in prospective trials to define extent of disease and to alter radiation treatment volumes.

18F-DCFPyL, a second generation PSMA PET agent that binds with high affinity to PSMA yet clears rapidly from the blood pool, has recently been approved by the FDA as a method to stage high risk cancer and detect recurrent disease.

Primary Objective:

To define 18F-DCFPyL PET/CT imaging response in participants with localized prostate cancer after treatment with stereotactic body radiation therapy (SBRT) with or without androgen deprivation therapy (ADT).

Eligibility:

Biopsy proven localized prostate cancer in whom prostate SBRT with or without ADT is appropriate therapy

Must have at least 1 MRI detected, biopsy proven site of prostate cancer.

ECOG 0-2

Design:

This is a single center, prospective study aimed at recruiting the following cohorts:

Up to 40 evaluable participants with presumed localized prostate cancer (intermediate or high risk) scheduled to undergo radiotherapy with systemic androgen deprivation therapy.

Up to 40 evaluable participants with presumed localized prostate cancer (intermediate or high risk) scheduled to undergo SBRT without androgen deprivation therapy.

Up to 20 evaluable participants with presumed localized prostate cancer (intermediate or high risk) scheduled to undergo radiotherapy with localized androgen deprivation therapy.

Participants receiving neoadjuvant androgen deprivation therapy will undergo a second 18F-DCFPyL PET/CT and multiparametric MRI (mpMRI) at 8 weeks after initiation of ADT but before SBRT.

All participants will undergo 18F-DCFPyL PET/CT and mpMRI 6 months following completion of SBRT and at recurrence, if applicable.

Participants will be followed for up to 2 years after completion of SBRT to evaluate longitudinal quality of life and biochemical control.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Biopsy proven localized prostate cancer in whom stereotactic body radiation treatment (SBRT) with or without neoadjuvant androgen deprivation therapy (ADT) is planned for definitive management (NIH laboratory of pathology confirmation is not required).
* Must have at least 1 MRI detected, biopsy proven localized prostate cancer.
* Age >= 18 years
* ECOG performance status <= 2
* For individuals with evidence of human immunodeficiency virus (HIV) infection, individuals must be on effective anti-retroviral therapy with undetectable viral load within the prior 6 months are eligible.
* For individuals with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* For individuals with a history of hepatitis C virus (HCV), the infection must have been treated and cured. For individuals with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Men must agree to use adequate contraception with their partner (hormonal or barrier method of birth control; abstinence) for the duration of study participation and 2 months after the last 18F-DCFPyL scan.

EXCLUSION CRITERIA:

* Receiving prior androgen deprivation therapy, radiotherapy, or surgery for prostate cancer.
* Any condition that is likely to interfere with study procedures or results.
* Individuals in whom pelvic nodal irradiation is planned.
* Serum creatinine > 2 times the upper limit of normal.
* Weighing > 350 lbs (weight limit for scanner table), or unable to fit in imaging gantry.
* Evidence of tumor spread beyond the prostate/seminal vesicles (lymph nodes, metastases).
* Contraindications to radiation or SBRT.

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Imaging response to treatment | Baseline, 8 weeks after ADT initiation (if applicable), 6 months post SBRT, at recurrence
  For the purpose of this study, the imaging response to treatment will be categorized separately in the radiation treatment volume (in field; local) and distantly (outside the radiation treatment volume). In-field (in the radiation target volume) 18F-DCFPyL PET/CT treatment response in field will be evaluated using a descriptor (complete, partial, progression) based on maximum SUV and volume of uptake relative to the pre-treatment imaging. Presence of new areas of uptake suspicious for prostate cancer outside of the region of radiation treatment will be considered progression but will be scored separately and will not impact the assessment of response from radiation locally.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000481-C.html